CLINICAL TRIAL: NCT00312676
Title: Conversion From Multiple-Daily Dose Enteric-Coated Depakote to Once-Daily Depakote ER in Elderly Outpatients With Epilepsy or Behavioral Disturbances:
Brief Title: Compare Tolerability of an Overnight Switch to Gradual Switch Between Two Different Forms of Depakote
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Veterans Affairs Medical Center, Miami (U.S. Federal Agency)
Collaborators: Abbott (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 7332.55b
Record Dates: First submitted 2006-04-06; First posted 2006-04-10 (Estimated); Last update posted 2006-04-10 (Estimated); Status verified 2006-03

CONDITIONS: Epilepsy; Behavioral Disturbance
Keywords: Tolerability; Depakote DR; Depakote ER; Elderly; Conversion
MeSH Terms: conditions — Epilepsy; Mental Disorders

INTERVENTIONS:
Procedure: Rapid versus slow conversion

SUMMARY:
The hypothesis is that the characteristics of extended release Depakote will allow overnight conversion of immediate release to extended release form of Depakote. This has been tested successfully in younger patients but not in individuals over the age of 60. We will include individuals between 60 and 80 years old.

DETAILED DESCRIPTION:
Twenty patients will be randomily assigned to convert overnight (10 pts) or over six days (10 pts). Side effects will be formally evaluated by the UKU side effect rating scal which will be done 7 days before conversion (day -7), the day of conversion (day 0)and then at the start of days +2, +7 and +14. This investigator conducting the evaluation will be blinded to the conversion status of the patient. Secondary measures to be obtained will be a Quality of Life measure (QOLIE-89) on Day 0 and +14. Plasma samples will be obtained on Day 0 and +14 before dosing for total and free valproic blood level.

ELIGIBILITY:
Inclusion Criteria:

* 60 yo and older on stable dose of valproate (Depakote DR)

Exclusion Criteria:

* Unstable neurolgical, medical or psychiatric disorder

Ages: 60 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20
Dates: Start 2006-03; Study Completion 2006-10

PRIMARY OUTCOMES:
Between group comparisons of GI and CNS side effect burden

SECONDARY OUTCOMES:
Between group comparison of Quality of Life as measured bye the QOLIE-89
Between group comparison of trough Total and Free valproic acid serum levels

CONTACTS AND LOCATIONS:
Overall Officials: R. Eugene Ramsay, MD, Principal Investigator — Miami Veterans Administration Medical Center
Locations (1):
- Miami VA Medical Center, Miami, Florida, United States